CLINICAL TRIAL: NCT06403488
Title: Letrozole Dose Increments in PCOS Patients Resistant to Letrozole Ovulation Induction
Brief Title: Letrozole Dose Increments in PCOS Patients Resistant to Letrozole
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Letrozole dose increments
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Letrozole; ovulation; PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- femara 1x3 (Experimental): Femara 2.5 mg (Novartis pharma ) 3 tablets per day starting from the second day of the menstrual cycle for 5 days
  Interventions: Drug: Letrozole 2.5mg
- femara 2x2 (Experimental): (Femara 2.5 mg (Novartis pharma )2 tablets twice daily for 5 days starting from the second day of the cycle
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Letrozole 2.5mg — specific aromatase inhibitor
  Other Names: femara

SUMMARY:
Objectives: To study the effect of Letrozole dose increments on ovulation rate and endometrial thickness as a primary outcomes in patients with polycystic ovary syndrome who previously resistant to letrazole conventional dose, and chemical and clinical pregnancy considered as secondary outcomes.

DETAILED DESCRIPTION:
A prospective cohort clinical trial study will be carried out at Beni Suef outpatient clinic from the period of October 2023 till January 2024, on 102 PCOS patients who received Letrozole for one month showing resistance or anovulation.

Inclusion criteria: Age 18 - 40 years old, normal semen analysis of their male partner, and diagnosis of PCOS based on a modified form of the Rotterdam criteria (at least two of the mentioned three criteria: chronic anovulation oligomenorrhea, clinical or biochemical signs of hyperandrogenism and polycystic ovaries on ultrasound).

Exclusion criteria: Any contraindications for pregnancy, and patients received other medications for ovulation induction such as metformin or clomiphene citrate and gonadotropins concomitantly, hyperprolactinemia; abnormal thyroid functions; multiple uterine fibroids; suspicion of endometriosis and adenomyosis The study performed on 102 PCOS patients resistant to conventional regimen for Letrozole, they were divided into 2 groups, Group A(received Femara 2.5 mg (Novartis pharma ) 3 tablets per day starting from the second day of the menstrual cycle for 5 days ) and Group B : received femara 2.5 mg (2 tablets twice daily for 5 days starting from the second day of the cycle. Transvaginal ultrasound for tracking follicular growth and endometrial thickness performed on 12th and 14th day of the cycle. Primary outcomes of the study were the follicular size and endometrial thickness (ovulation detection). Secondary outcomes were the biochemical and clinical pregnancy rates.

Ethical considerations Approval by the institution ethical committee, The Beni-Suef University Faculty of Medicine Research Ethics Committee has approved the study (FMBSUREC/03102023/Ali). Individual consent process: informed consent was taken after explaining the study objectives and procedures to each patient.

Sample size was calculated using G*power (8) for sample size calculation, based on assumption that effect size was 0.5. For a confidence 95% and power 80%, and assumption for using a t-test for two independent means groups, the minimum required sample size is 102 participants with 51 participants in each group.

Data analysis and statistics Categorical data were reported as numbers and proportions and comparisons were performed using chi-square and the Fisher exact test when appropriate. Continuous variables were presented using mean and standard deviation and compared using an unpaired t-test for normally distributed data and Mann-Whitney U test for data was not normally distributed. A value of p < 0.05 was considered statistically significant. All statistical analyses were performed with Statistical Package for Social Sciences (SPSS), version 26 (SPSS Inc., Chicago, IL, USA)

ELIGIBILITY:
Inclusion Criteria:

* normal semen analysis of their male partner
* Diagnosis of PCOS based on a modified form of the Rotterdam criteria

Exclusion Criteria:

* Any contraindications for pregnancy
* patients received other medications for ovulation induction such as metformin or clomiphene citrate and gonadotropins concomitantly
* hyperprolactinemia
* abnormal thyroid functions
* multiple uterine fibroids

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 1 month
  the follicular size by trans-vaginal ultrasound reached more than 18 mm
endometrial thickness | 1 cycle (1month)
  assessed by trans-vaginal ultrasound

SECONDARY OUTCOMES:
pregnancy rate | 1 month
  positive HCG test

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate
  - Beni-suef university Hospital, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No